CLINICAL TRIAL: NCT01758679
Title: A Clinical Trail of Iodine[131I] Metuximab Injection With CIK Cells for Preventing Relapse and Metastasis of Hepatocellular Carcinoma
Brief Title: A Clinical Trail of Iodine[131I] Metuximab Injection With CIK Cells for Preventing Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIH-XWG-201205001
Record Dates: First submitted 2012-08-29; First posted 2013-01-01 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2012-08

CONDITIONS: Multiple Drug Use
Keywords: Iodine[131I] Metuximab Injection
MeSH Terms: interventions — metuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Licartin，Licartin and CIK (Experimental): Intravenous Licartin 27.75 M Bq(0.75 mCi)/kg Licartin and CIK
  Interventions: Biological: Licartin and CIK

INTERVENTIONS:
Biological: Licartin and CIK — Licartin and CIK

SUMMARY:
This clinical trial is designed to provide one kind of modalities for preventing the recurrence and metastasis of PLC. If the expected therapeutic efficacy is achieved, it shall contribute actively to boosting the therapeutic level of PLC, prolonging its recurrent time and enhancing its overall survival. And it may also raise the clinical recognition of this technology, promote its clinical applications and generate excellent social reputations and economic returns.

DETAILED DESCRIPTION:
Primary liver cancer (hereinafter abbreviated as PLC) is one of the most common types of malignant tumors in clinical practices. Its global prevalence is rising year-on-year and surpasses 626,000 per year. Ranking at No. 5 among all malignant tumors, its mortality rate approaches 600,000 per year and becomes No.3 of tumor-related death. As one of the prevalent regions of PLC in the world, China has a morbidity population of around 55%. Among the tumor-related death, it stands at No. 2 second only to lung cancer. So PLC has been a major hazard to health and life for Chinese citizens. Surgical resection has remained the first therapeutic choice of PLC. However, the disease course of PLC is insidious. In clinical practices, less than 30% of PLC patients may be treated surgically by hepatectomy. And their postoperative occurrences of recurrence and metastasis stay at a high level. As demonstrated by large-sample clinical trials in China, the 5-year postoperative recurrent rate of PLC was as high as 61.5%. The relevant studies have indicated that the surgical therapy of PLC has encountered a bottle-neck over the last decade and the control rates of postoperative recurrence or metastasis remain basically the same. Therefore the recurrence and metastasis of PLC are important limiting factors for its clinical therapeutic gains. Effectively lowering the post-therapeutic recurrence and metastasis of PLC has become a breakthrough point for improved clinical efficacies. At present, there is still no standard therapeutic protocol for the prevention of recurrence and metastasis of PLC.

Independently developed recently by China, licartin has been the first radioimmunological targeted therapeutic agent approved for PLC in the world. Since its marketing in 2007, it has achieved excellent clinical efficacies and social recognition. As demonstrated by the results of relevant basic and clinical researches, licartin had definite efficacies for primary hepatocellular carcinoma and it could boost the efficacies of integrated PLC therapy, prolong the patient survivals and enhance the benefits of clinical therapeutics. Early studies have also proved that it could prolong the survivals of PLC, improve the quality of life and prevent the postoperative recurrence and metastasis. The present clinical trial is intended to examine the efficacy and safety of radioimmunotherapy via intravenous infusion of licartin plus sequential immunotherapy of CIK cell in the controls of disease progression, effective prolonging of recurrent time and prevention of recurrence or metastasis of primary hepatocellular carcinoma.

This clinical trial is designed to provide one kind of modalities for preventing the recurrence and metastasis of PLC. If the expected therapeutic efficacy is achieved, it shall contribute actively to boosting the therapeutic level of PLC, prolonging its recurrent time and enhancing its overall survival. And it may also raise the clinical recognition of this technology, promote its clinical applications and generate excellent social reputations and economic returns.

ELIGIBILITY:
Inclusion Criteria:

* Definite pathological diagnosis of hepatocellular carcinoma
* Excellent healing of surgical wounds, no overt surgical complication and stable disease
* Such imaging examinations as ultrasound, CT and MRI reveal no definite tumor foci
* Subject's physical status:Karnofsky performance status score ≥70 points
* Metuxitab skin test negative
* Receiving no radiotherapy, chemotherapy or molecular targeted therapy within 4 weeks pre-therapy
* Male/female aged 18-70 years
* Expected survival period > 3 months
* Voluntary group participation, excellent compliance, cooperative in observations and signing a written informed consent form.

Exclusion Criteria:

* Poor general constitution with obviously impaired liver function (bilirubin > 3 folds of normal upper limit and serum albumin <30 g/L)
* Blood routine examination: white blood cell <4.0×109/L or platelet count <80×109/L
* Definite tumor foci found on such imaging examinations of ultrasound, CT or MRI
* Postoperative onset of recurrence or metastasis and no clinical remission after therapy
* Severe infection, such as hepatic abscess
* Abnormal thyroid functions
* Obvious cases of pleural effusion and ascites
* Diffuse systemic metastasis and therapy is not expected to prolong the patient's survival period
* Poor compliance
* Patients with a history of hypersensitivity to biological preparations, hypersensitive physique or currently in a hypersensitive state
* Pregnant and lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhao, Doctor, Study Director — Director of Pharmacology Base
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China